CLINICAL TRIAL: NCT03354715
Title: Patient Satisfaction and Retention of Upper Complete Denture Base Using Rapid Prototyping Versus a Conventional One: Randomized Control Trial
Brief Title: Patient Satisfaction and Retention of Upper Complete Denture Base Using Rapid Prototyping Versus a Conventional One
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Mahmoud Youssef, Master Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2717
Record Dates: First submitted 2017-07-30; First posted 2017-11-28 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Complete Denture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid prototyping Denture base (Sham Comparator): Complete Denture Using Rapid Prototyping method for fabrication of the complete denture depending on
  Interventions: Device: Rapid prototyping Denture base
- Heat Cured Conventional Complete Denture (Sham Comparator): Complete Denture using heat cured Denture base using flasking and deflasking method
  Interventions: Device: Heat Cured Conventional Complete Denture

INTERVENTIONS:
Device: Rapid prototyping Denture base — The introduction of rapid prototyping (RP)Stereo lithography (SLA) technology, which mainly depends on addition of layers of materials which would be polymerized using a light curing unit. It consists of a bath of photo polymerized liquid and ultraviolet unit for curing these layers, that would bond to each other till forming the full object. SLA has many advantage as high accuracy, high mechanical strength, smooth surface finish with close tolerance and fine details printing, but it has some limitation as it is only limited Material, in addition to the high material and equipment cost.
  Arms: Rapid prototyping Denture base
Device: Heat Cured Conventional Complete Denture — it is the main treatment for most of completely edentoulous Cases
  Arms: Heat Cured Conventional Complete Denture

SUMMARY:
Comparing patient satisfaction and retention of upper complete denture fabricated using two different denture base materials, the first fabricated using rapid prototyping method while the second is following conventional methods.

DETAILED DESCRIPTION:
Searching for other materials or other fabrication technologies has been one of the goals to help to re-innovate the fabrication of complete dentures , which would greatly influence completely edentulous Patient satisfaction. The introduction of rapid prototyping (RP)Stereo lithography (SLA) technology has many advantage as high accuracy, high mechanical strength, smooth surface finish with close tolerance and fine details printing, but it has some limitation as it is only limited Material, in addition to the high material and equipment cost.

SLA has been used in dental fields like maxillofacial prosthesis , wax pattern fabrication for crown bridge , removable partial denture 19, but still complete denture was reported in a very few reports indicating that RP is not yet successfully applied in Complete denture manufacturing 19-21A randomised trial is therefore needed to asses accurately wether the introduction of rapid prototyping in complete denture fabrication is successful or not in comparison to the conventional technique and to discover the possible challenges in this recent technique and the ways to overcome it.

Retention of complete dentures and patient satisfaction has been reported in many studies22-26. Patients have showed a higher satisfaction, as retention of both maxillary and mandibular complete dentures increased.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 40-70 years.
2. Patients who can understand and respond to a written questionnaire in Arabic.
3. Cooperative patients

Exclusion Criteria:

1. Pathological changes of residual ridges.
2. Patients with debilitating systemic diseases.
3. Patients with xerostomia.
4. Patients with flabby and flat ridges.
5. Patients with allergy to acrylic resin
6. Patient with sever undercuts, or irregular bony exostosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 3 month
  Patient Satisfaction Questionnaire using likert scale five points represent degree of satisfaction and compare the result to each other

SECONDARY OUTCOMES:
Retention | 3 month
  resistance to tissue away movement using digital force meter and recording the average of 10 reading in one time and compare the results of the two denture

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided